CLINICAL TRIAL: NCT03531255
Title: An Open Label, Non-Randomized, Multi-Center Extension Study to Evaluate the Long-Term Safety and Efficacy of Pegcetacoplan in the Treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Pegcetacoplan Long Term Safety and Efficacy Extension Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-307
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: PNH
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1,080 mg pegcetacoplan administered subcutaneously (Experimental): 1,080mg pegcetacoplan administered subcutaneously twice weekly or every three days.
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor

SUMMARY:
This is an Open-label, Non-Randomized, Multi-Center Extension Study. Eligible subjects will have previously completed a pegcetacoplan study.

ELIGIBILITY:
Inclusion criteria:

1. Subjects at least 18 years of age with PNH who have participated in a pegcetacoplan clinical trial. Subjects who received treatment with pegcetacoplan must have experienced clinical benefit and adequate tolerability in the opinion of the investigator.

   Note: Subjects with PNH who completed a pegcetacoplan clinical trial without receiving pegcetacoplan (or without receiving pegcetacoplan for long enough to demonstrate clinical benefit) may be enrolled in this study if, in the opinion of the Investigator, the subject is expected to demonstrate clinical benefit upon the initiation or continuation of pegcetacoplan therapy.
2. Vaccination against Neisseria meningitidis types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) either within 2 years prior to Day 1 dosing of this study, or within 14 days after starting treatment with pegcetacoplan. Vaccination is mandatory unless documented evidence exists that subjects are nonresponders to vaccination as evidenced by titers or display titer levels within acceptable local limits. Immunization status checks will be performed to determine whether subjects require primary or booster vaccinations.
3. Willing and able to give written informed consent.
4. Willing and able to self-administer pegcetacoplan (administration by caregiver will be allowed)
5. Women of childbearing potential (WOCBP) defined as any females who have experienced menarche and who are NOT permanently sterile or postmenopausal must have a negative pregnancy test and must agree to continue to use an approved method of contraception for the duration of the study and 90 days after their last dose of study drug. Note: Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.
6. Males must agree to continue to use an approved method of contraception and must agree to refrain from donating sperm for the duration of the study and 90 days after their last dose of study drug.

Exclusion Criteria:

1. Subjects who have withdrawn from a pegcetacoplan clinical study.
2. Any condition that could increase the subject's risk by participating in the study.
3. Any comorbidity or condition (such as malignancy) that, in the opinion of the investigator, could put the subject at increased risk or potentially confound study data.
4. History or presence of hypersensitivity or idiosyncratic reaction to compounds related to the investigational product or SC administration.
5. Known infection with hepatitis B, C, or HIV.
6. Hereditary complement deficiency.
7. History of bone marrow transplant.
8. Concurrent severe aplastic anemia (SAA), defined as currently receiving immunosuppressive therapy for SAA including but not limited to cyclosporin A, tacrolimus, mycophenolate mofetil or anti-thymocyte globulin.
9. History of meningococcal disease.
10. Concomitant treatment with any complement inhibitor (eg, eculizumab, ravulizumab).
11. Pregnancy, breastfeeding, or positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Baseline to 2 Years

CONTACTS AND LOCATIONS:
Locations (62):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Denver Health Medical Center, Denver, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Lakes Research, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Baptist Cancer Center, Memphis, Tennessee
- Royal Melbourne Hospital, Melbourne, Victoria, Australia
- Belgium (2):
  - Cliniques Universitaires Saint-luc, Brussels
  - AZ Delta, Roeselare
- Bulgaria (2):
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - National Specialized Hospital for Active Treatment of Haematologic Diseases, Sofia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
- IPS Centro Medico Julian Coronel SAS, Cali, Valle del Cauca Department, Colombia
- France (6):
  - Hospital Center Chalon Sur Saone William Morey, Chalon-sur-Saône
  - CHRU de Lille, Lille
  - Hopital Saint-Louis, Paris
  - Lyon Sud Hospital Center, Pierre-Bénite
  - Centre Hospitalier Annecy Genevois - Site Annecy, Pringy
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
- Germany (4):
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Essen University Hospital Department of Hematology, Essen, North Rhine-Westphalia
  - University Medical Center Hamburg-Eppendorf, Hamburg
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Japan (6):
  - Japanese Red Cross Nagoya Daini Hospital, Showa-ku, Aichi-ken
  - Shinshu University Hospital, Matsumoto, Nagano
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - Kinan Hospital, Tanabe, Wakayama
  - Okayama University Hospital, Okayama
  - NTT Medical Center Tokyo, Tokyo
- Malaysia (2):
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Ampang, Ampang, Selangor
- Hospital Universitario "José Eleuterio González", UANL, Monterrey, Mexico
- Peru (3):
  - Hospital Nacional Dos De Mayo - Centro de Investigación, Lima Cercado, Lima region
  - Centro de Investigacion en Hematologia Clinica del Centro Medico Corpac, San Isidro, Lima region
  - Hospital Edgardo Rebagliatti, Jesús María, Lima
- Philippines (5):
  - Perpetual Succour Hospital, Cebu, National Capital Region
  - Mary Mediatrix Medical Centre, Lipa City, National Capital Region
  - Makati Medical Centre, Makati City, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - St. Lukes Medical Centre, Quezon City, National Capital Region
- Russia (2):
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Therapeutic hospital of regional clinical hospital #1, Tyumen
- Clinical Center of Serbia, Belgrade, Serbia
- Singapore General Hospital, Singapore, Singapore
- Chungnam National University Hospital, Junggu, Daejeon, South Korea
- Spain (2):
  - Hospital Univ. de Gran Canaria Dr.Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Politecnico La Fe, Valencia
- Thailand (7):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Songklanagarind Hospital, Songkhla
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Derived] de Castro C, Kelly RJ, Griffin M, Patriquin CJ, Mulherin B, Hochsmann B, Selvaratnam V, Wong RSM, Hillmen P, Horneff R, Uchendu UO, Zhang Y, Surova E, Szamosi J, de Latour RP. Efficacy and Safety Maintained up to 3 Years in Adults with Paroxysmal Nocturnal Hemoglobinuria Receiving Pegcetacoplan. Adv Ther. 2025 Sep;42(9):4641-4658. doi: 10.1007/s12325-025-03310-8. Epub 2025 Jul 28. PMID 40720060
- [Derived] Patriquin CJ, Bogdanovic A, Griffin M, Kelly RJ, Maciejewski JP, Mulherin B, Peffault de Latour R, Roth A, Selvaratnam V, Szer J, Al-Adhami M, Horneff R, Tan L, Yeh M, Panse J. Safety and Efficacy of Pegcetacoplan in Adult Patients with Paroxysmal Nocturnal Hemoglobinuria over 48 Weeks: 307 Open-Label Extension Study. Adv Ther. 2024 May;41(5):2050-2069. doi: 10.1007/s12325-024-02827-8. Epub 2024 Apr 4. PMID 38573482
- [Derived] Griffin M, Kelly RJ, Panse J, de Castro C, Szer J, Horneff R, Tan L, Yeh M, Peffault de Latour R. Management of acute breakthrough hemolysis with intensive pegcetacoplan dosing in patients with PNH. Blood Adv. 2024 Apr 9;8(7):1776-1786. doi: 10.1182/bloodadvances.2023011691. PMID 38315872
- [Derived] Sharma V, Koprivnikar J, Drago K, Savage J, Bachelor A. Injection Site Reactions with Long-Term Pegcetacoplan Use in Patients with Paroxysmal Nocturnal Hemoglobinuria: A Brief Report. Adv Ther. 2023 Nov;40(11):5115-5129. doi: 10.1007/s12325-023-02653-4. Epub 2023 Sep 14. PMID 37707673